CLINICAL TRIAL: NCT00847392
Title: Pediatric Volumetric Bladder Ultrasound Study
Brief Title: Study to Determine Pediatric Bladder Volume Prior to Catheterization
Acronym: PV-BUS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to obtain grant funding
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Dr. Andrew Worster, Hamilton Health Sciences
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PV-BUS
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Urinary Tract Infection
Keywords: Urethral catheterization; Emergency Department; Ultrasound; Urinary tract infection; Pediatric
MeSH Terms: conditions — Urinary Tract Infections; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound (Experimental): Bladder ultrasound prior to catheterization
  Interventions: Procedure: Ultrasound prior to bladder catheterization
- Standard catheterization (No Intervention): No ultrasound prior to bladder catheterization

INTERVENTIONS:
Procedure: Ultrasound prior to bladder catheterization — Bedside ultrasound to estimated volume of urine in bladder
  Arms: Ultrasound

SUMMARY:
This is a randomized controlled trial evaluating the effectiveness of bedside volumetric bladder ultrasound prior to transurethral catheterization of pediatric patients presenting to an emergency department with suspected urinary tract infection.

Ultrasound prior to catheterization allows Emergency Physicians to determine if the urine volume of the bladder is sufficient for successful catheterization. Advance knowledge of insufficient urine allows the Emergency Physician to defer the procedure until success is likely.

ELIGIBILITY:
Inclusion Criteria:

* Children 0-36 months of age
* Require urethral catheterization for urine analysis

Exclusion Criteria:

* Recently voided and unlikely to provide sufficient urine when catheterized
* Documented or suspected genitourinary abnormalities precluding urethral catheterization
* Indwelling catheter or urostomy
* Critical illness
* No available legal guardian or legal guardian does not understand English well enough to provide informed consent
* Technical failure of the utlrasound equipment

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients in each arm from whom at least 2 ml of urine is obtained on first attempt at catheterization. | First feasible attempt at catheterization during ED visit (minutes-hours).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Worster, MD, MSc, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada